CLINICAL TRIAL: NCT02035176
Title: Oregon Animation Test for Social Reciprocity (OATS)
Brief Title: Novel Measure of Social Deficits in Children
Acronym: OATS
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Garet Lahvis, Assistant Professor, Oregon Health and Science University
Other Study IDs: eIRB 9747
Record Dates: First submitted 2013-11-06; First posted 2014-01-14 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorders; ADHD
Keywords: autism; ADHD; attention deficit hyperactivity disorder; behavioral assessment; behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Autistic children ages 6-11: Autistic children ages 6-11
- ADHD children ages 6-11: ADHD children ages 6-11
- Typical children ages 6-11: Typical children ages 6-11

SUMMARY:
Autism Spectrum Disorders (ASD) feature impairments in social interaction and communication. Drug and behavioral treatments for ASD are undergoing rapid development, yet our diagnostic tools are not suitable for efficacy assessment. The Autism-Diagnosis Observational Schedule (ADOS) is a clinical interview with the child and the gold standard for diagnosis. However, this test is subjective, course grained and costly, precluding repeated tests of the same child to assess treatment efficacy and large-scale control assessments of typically developing (TD) children. For these reasons, the ADOS can impede imaging and genetic research.

In light of these concerns, the Oregon Animation Test for Social Reciprocity (OATS) will be developed to evaluate distinct autistic behavioral phenotypes, including joint attention, empathy, imitation, and lack of narrative coherence. The main idea of OATS is that animated characters and social scenarios are presented on a computer screen while the responses of the child are recorded by video camera, microphone, and eye-tracking equipment. Animations are used to test each behavioral phenotype of autism. The long-term vision for OATS is to evaluate behavioral and physiological responses of autistic children, including heart rate variability, pupil dilation, and EEG. Our first objective is to use existing animations to build an OATS "Prototype" that discriminates autistic from normal children (Aim 1). From these results, and use of a defined library of still frame posed images, we will design our own animation platform to assess differences between autistic and normal children (Aim 2).

DETAILED DESCRIPTION:
Please see the brief summary above.

ELIGIBILITY:
Inclusion Criteria:

* 6-11 years of age with autism,
* ADHD, or typical

Exclusion Criteria:

* IQ below 70.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 6-11 years of age with autism, ADHD, or typical, with and IQ exceeding 70.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2014-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Eye gaze in response to animated social situations | 60 minutes

SECONDARY OUTCOMES:
Facial expressions in response to animated social situations | 60 minutes
  A child is shown an animation and facial expressions are coded for various emotions.

OTHER OUTCOMES:
Ability to recount a story shown via animation | 10 minutes
  A child is shown an animation and is asked to recount the story.
Ability to imitate an action shown via animation | 10 minutes
  A child is shown an animation and is asked to imitate a character's action .

CONTACTS AND LOCATIONS:
Overall Officials: Garet P Lahvis, PhD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - OHSU, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon